CLINICAL TRIAL: NCT01928693
Title: A Single-site, Single Masked, Prospective Comparison of Three Fluoroquinolone Topical Therapies (Besifloxacin 0.6% or Gatifloxacin 0.5% or Moxifloxacin 0.5%) in the Treatment of Infectious Corneal Ulcers.
Brief Title: A Comparison of Three Fluoroquinolone Topical Eyedrops in the Treatment of Infectious Corneal Ulcers.
Acronym: Eye02
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study terminated due to slow accrual
Sponsor: Cornea Consultants Of Nashville (Other)
Collaborators: SCRI Development Innovations, LLC (Other); Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eye02
Record Dates: First submitted 2013-08-20; First posted 2013-08-27 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Corneal Ulcers
Keywords: infectious corneal ulcers
MeSH Terms: conditions — Corneal Ulcer | interventions — besifloxacin; Gatifloxacin; Ophthalmic Solutions; Moxifloxacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Besivance 0.6% Ophthalmic Suspension (Active Comparator): A topical fluoroquinolone antimicrobial indicated for the treatment of bacterial conjunctivitis.
  Interventions: Drug: Besivance 0.6% Ophthalmic Suspension
- Zymaxid 0.5% Ophthalmic Solution (Active Comparator): A topical fluoroquinolone anti-infective indicated for the treatment of bacterial conjunctivitis.
  Interventions: Drug: Zymaxid 0.5% Ophthalmic Solution
- Vigamox 0.5% Ophthalmic Solution (Active Comparator): A topical fluoroquinolone anti-infective indicated for the treatment of bacterial conjunctivitis.
  Interventions: Drug: Vigamox 0.5% Ophthalmic Solution

INTERVENTIONS:
Drug: Besivance 0.6% Ophthalmic Suspension — Drop to be applied in affected eye initially every hour for the first 48 hours then doses will be reduced at each subsequent visit by 50% if patient continues to show a reduction in size of 25% from the previous visit up to every 4 hours. If subject dose has been reduced to every 4 hours at visit 3 and shows an additional reduction size of 25% at visit 4, then they will be reduced to every 6 hours.
  Other Names: Besifloxacin 0.6% Ophthalmic Suspension
  Arms: Besivance 0.6% Ophthalmic Suspension
Drug: Zymaxid 0.5% Ophthalmic Solution — Drop to be applied in affected eye initially every hour for the first 48 hours then doses will be reduced at each subsequent visit by 50% if patient continues to show a reduction in size of 25% from the previous visit up to every 4 hours. If subject dose has been reduced to every 4 hours at visit 3 and shows an additional reduction size of 25% at visit 4, then they will be reduced to every 6 hours.
  Other Names: Gatifloxacin 0.5% Ophthalmic Solution
  Arms: Zymaxid 0.5% Ophthalmic Solution
Drug: Vigamox 0.5% Ophthalmic Solution — Drop to be applied in affected eye initially every hour for the first 48 hours then doses will be reduced at each subsequent visit by 50% if patient continues to show a reduction in size of 25% from the previous visit up to every 4 hours. If subject dose has been reduced to every 4 hours at visit 3 and shows an additional reduction size of 25% at visit 4, then they will be reduced to every 6 hours.
  Other Names: Moxifloxacin Hydrochloride 0.5% Ophthalmic Solution
  Arms: Vigamox 0.5% Ophthalmic Solution

SUMMARY:
This Phase II study will evaluate the safety and efficacy of three fluoroquinolone ophthalmic agents to determine the optimal treatment in patients with infectious corneal ulcers.

DETAILED DESCRIPTION:
This is a prospective, single masked, comparative, mono-therapeutic trial evaluating three fluoroquinolone agents that are approved and marketed for the treatment of conjunctivitis. Approximately 120 patients who have corneal ulcers greater than 2 mm but less than 6 mm in size who meet all other inclusion criteria will be enrolled into this study. Patients will be randomized in a 2:1:1 ratio to receive besifloxacin 0.6% ophthalmic suspension, gatifloxacin 0.5% ophthalmic solution, or moxifloxacin 0.5% ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be between the ages of 18-90 years of age.
2. Patients must be able to understand the nature of this study, give written informed consent prior to study entry, and comply with study requirements.
3. Patients must have a corneal ulcer greater than 2mm but less than 6mm in size.
4. Patients must have corneal ulcer present in only one eye.
5. Patients must agree not to wear contact lenses while on study.

Exclusion Criteria:

1. Patients with multifocal ulcers.
2. Signs of any other viral or fungal infection.
3. Treatment with antibiotics within 14 days of study entry.
4. Treatment with systemic or topical ocular antiviral agents or systemic or topical steroids or topical ocular nonsteroidal anti-inflammatory drugs (NSAIDS) during the prior 14-day period.
5. Known hypersensitivity or allergy to steroids (Loteprednol etabonate) or to any of the ingredients in the three study drugs (Besifloxacin 0.6% or Gatifloxacin 0.5% or Moxifloxacin 0.5%).
6. Contact lens only with no spectacles available.
7. Ocular surgery (including laser surgery) in either eye within 6 weeks prior to entry into this study.
8. Participation in any investigational study within the past 30 days.
9. Pregnant women, minors, or those not able to consent for themselves.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira A. Shivitz, M.D., Principal Investigator — Cornea Consultants Of Nashville
Locations (1):
- Cornea Consultants of Nashville, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Started | 0 | 1 | 1
Completed | 0 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution | Total
Number analyzed (Participants) | 0 | 1 | 1 | 2
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0 | 0
  Between 18 and 65 years |  | 0 | 1 | 1
  >=65 years |  | 1 | 0 | 1
Gender [Number; unit: participants]
  Female |  | 1 | 0 | 1
  Male |  | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Healing
Description: The primary outcome will be complete healing of the corneal ulcer, defined as complete reepithelialization by Day 29.
Time Frame: 29 days
Measure: Number; unit: participant
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Number analyzed (Participants) | 0 | 1 | 1
participant |  | 1 | 1

2. Secondary Outcome: Healing Rate
Description: Time to corneal ulcer reduction and/or total healing over a treatment course of 21 days.
Time Frame: 29 days
Measure: Number; unit: Days
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Number analyzed (Participants) | 0 | 1 | 1
Days |  | 21 | 21

3. Other Pre Specified Outcome: Time to Treatment Failure.
Description: If there is no reduction in size of the corneal ulcer by day 8, the treatment will be deemed a failure and alternative medications will be given at the discretion of the investigator.
Time Frame: 8 days
Population: Data was not collected because there were no treatment failures in any of the treatment arms
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Scarring
Description: Scarring will be evaluated and measured in millimeters at Day 29 and classified as either peripheral or central.
Time Frame: 29 days
Measure: Number; unit: millimeters
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Number analyzed (Participants) | 0 | 1 | 1
millimeters |  | 0 | 0

5. Other Pre Specified Outcome: Patient Satisfaction Scores
Description: Patient satisfaction outcomes will be assessed using a series of survey questions ranging in both categorical and continuous outcomes. Treatment will be compared using either methods for differences in binomial proportions or the Wilcoxon Rank Sum test. Scale= 0- Very Comfortable, 1- Comfortable, 2- Uncomfortable, 3- Very Uncomfortable
Time Frame: Average of 6 times in a 29 day period
Measure: Number; unit: units on a scale
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Number analyzed (Participants) | 0 | 1 | 1
units on a scale |  | 0 | 2

6. Other Pre Specified Outcome: Patient Pain Scores
Description: Patients will be asked to grade the overall pain of the affected eye at each visit on a Scale= 0--None, 1- Mild, 2- Moderate, 3- Severe
Time Frame: Average of 6 times in a 29 day period
Measure: Number; unit: units on a scale
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Number analyzed (Participants) | 0 | 1 | 1
units on a scale |  | 0 | 2

7. Other Pre Specified Outcome: Number of Participants With Treatment Failure
Time Frame: 29 days
Measure: Number; unit: participants
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Number analyzed (Participants) | 0 | 1 | 1
participants |  | 0 | 0

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | Besivance 0.6% Ophthalmic Suspension | Zymaxid 0.5% Ophthalmic Solution | Vigamox 0.5% Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes